CLINICAL TRIAL: NCT06292598
Title: Bacterial Translocation and Gut Microbiota in Type 1 Narcolepsy Patients
Brief Title: Bacterial Translocation and Gut Microbiota in Type 1 Narcolepsy Patients Versus a Control Population
Acronym: NARCOBIOTE
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: AOI2022/2023/CDR-01
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Narcolepsy Type 1; Bacterial Translocation
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and fecal samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with untreated NT1
  Interventions: Other: Blood sample; Other: Stool sample; Other: CSF sample
- Matched controls: Controls matched on sex, age (+/- 2 years) and BMI class (BMI < 25: normal; 25 ≤ BMI ≤ 30: overweight; BMI > 30: obesity)
  Interventions: Other: Blood sample; Other: Stool sample

INTERVENTIONS:
Other: Blood sample — Sample taken to test plasma permeability markers
Other: Stool sample — Sample taken to test microbial diversity and composition
Other: CSF sample — Sample taken to test orexin level
  Groups: Patients with untreated NT1

SUMMARY:
Narcolepsy type 1 (NT1) is a rare disease characterized by severe drowsiness, cataplexy, hypnagogic hallucinations, sleep paralysis, poor night sleep, and often obesity. NT1 is caused by irreversible loss of orexin (ORX)/hypocretin neurons in the lateral hypothalamus with decreased ORX levels in the cerebrospinal fluid (CSF). Although the underlying process leading to this destruction remains unclear; an autoimmune origin is suspected.

The study authors recently compared the bacterial communities of the fecal microbiota of NT1 patients and control subjects. Initial results demonstrated a difference in overall bacterial community structure in NT1 compared to controls, as assessed by beta diversity, even after adjusting for body mass index (BMI). The Shannon biodiversity index was also correlated with the duration of NT1 disease. However, no association was found between the structure of the microbial community and the clinical characteristics of NT1 patients.

In 2022, a second study from the SOMNOBANK cohort on a larger population confirmed these results, showing dysbiosis between NT1 patients and the control population. The altered intestinal microbial diversity supports the important role of the environment in the development and pathogenesis of NT1. Other studies have established a link between dysbiosis, intestinal permeability and inflammation in other neuroimmune pathologies. Currently, no study has focused on these phenomena of bacterial translocation, intestinal permeability and immune activation linked to the microbiota in type 1 narcolepsy patients.

The study hypothesis is that NT1 patients with dysbiosis in their intestinal microbiota also present a bacterial translocation with an intestinal origin, leading to a systemic inflammatory syndrome favoring an autoimmune damage destroying hypocretin neurons in the hypothalamus. The study authors suspect that microbial elements (DNA) involved in the autoimmune process could be detected in the CSF. This bacterial translocation could vary over time depending on: i) the progression of the disease and its management; ii) changing dysbiosis and: iii) the increase in intestinal permeability and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with narcolepsy type 1 (NT1).
* Patient not treated for narcolepsy during initial evaluation of NT1 patients.
* Patient eligible for treatment for longitudinal monitoring of NT1 patients.
* Patient speaking and understanding French.
* The patient must have given their free and informed consent and signed the consent form or consent has been provided from the holder(s) of parental authority or the legal guardian and the child.
* The patient must be a member or beneficiary of a health insurance plan

Inclusion criteria for control subjects:

• Absence of diagnosis of sleep disorder responsible for hypersomnolence with an Epworth sleepiness scale score greater than 10/24.

Exclusion Criteria:

* Subject having presented an infectious pathology requiring antibiotic treatment in the previous 3 months.
* Subject with a dysimmune pathology.
* Subject having had treatment with an immunomodulatory molecule or chemotherapy within 60 days before inclusion in the research or whose indication is planned for the duration of the research.
* Subject with a chronic digestive pathology or having undergone bariatric surgery in the previous year.
* Subject on laxative.
* Subject living in a medical institution.
* Subject under legal protection, guardianship or curatorship.
* Subject and/or their legal representative (if a minor patient) unable to express consent
* Taking antibiotics during the inclusion period, or laxative or any other treatment having a significant impact on the microbiota

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults or children (≥10 years) with type 1 narcolepsy managed at the Montpellier and Nîmes teaching hospitals. This population will be matched on sex, age (± 2 years) and BMI class (BMI < 25: normal; 25 ≤ BMI ≤ 30: overweight; BMI > 30: obese) with a population of control subjects without central hypersomnolence, consulting the participating services mainly for another sleep disorder.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Plasma bacterial translocation profiles between groups | Day 0
  Circulating plasma r16s DNA (copies/μL)

SECONDARY OUTCOMES:
Plasma bacterial translocation profiles in NT1 patients | Month 12
  Circulating plasma r16s DNA (copies/μL)
Taxonomic characteristics of DNA in the CSF of NT1 patients according to narcolepsy severity | Day 0
  Metagenomic sequencing of all genomes present, compared with international databases, presented as number of reads per species (bacterial, fungal and viral)
Taxonomic characteristics of plasma bacterial DNA in patients with high bacterial translocation | Day 0
  Metabarcoding of 16srDNA of bacterial DNA present in plasma in NT1 patients with 16S rDNA >25 copies/μL, presented as relative abundance of bacterial phyla and genera (%)
Taxonomic characteristics of plasma bacterial DNA in patients with high bacterial translocation | Month 12
  Metabarcoding of 16srDNA of bacterial DNA present in plasma in NT1 patients with 16S rDNA >25 copies/μL, presented as relative abundance of bacterial phyla and genera (%)
Beta diversity of the intestinal microbiota between groups | Day 0
  measured by metabarcoding
Beta diversity of the intestinal microbiota in NT1 patients | Month 12
  measured by metabarcoding
Alpha diversity of the intestinal microbiota between groups | Day 0
  measured by metabarcoding
Alpha diversity of the intestinal microbiota in NT1 patients | Month 12
  measured by metabarcoding
Composition of the intestinal microbiota between groups | Day 0
  Relative abundance of bacterial phyla and genera (%) measured by metabarcoding
Composition of the intestinal microbiota between groups | Month 12
  Relative abundance of bacterial phyla and genera (%) measured by metabarcoding
Plasma Intestinal Fatty Acid Binding Protein (i-FABP) profile between groups | Day 0
  Measured by ELISA (pg/mL)
Plasma Intestinal Fatty Acid Binding Protein (i-FABP) profile in NT1 patients | Month 12
  Measured by ELISA (pg/mL)
Plasma LPS-binding Protein (LBP) profile between groups | Day 0
  Measured by ELISA (μg/mL
Plasma LPS-binding Protein (LBP) profile in NT1 patients | Month 12
  Measured by ELISA (μg/mL
Plasma Soluble CD14 profile between groups | Day 0
  Measured by ELISA (μg/mL
Plasma Soluble CD14 profile in NT1 patients | Month 12
  Measured by ELISA (μg/mL
Age of onset of symptoms in NT1 patients | Day 0
  Years
Duration of disease progression in NT1 patients | Day 0
  Years
Severity of sleep-related symptoms in NT1 patients | Day 0
  Epworth scale
Severity of narcolepsy symptoms in NT1 patients | Day 0
  Narcolepsy Severity Scale
Description of comorbidities in NT1 patients | Day 0
  List
Sleep onset latency in NT1 patients | Day 0
  Minutes
Number of rapid eye movement sleep episodes in NT1 patients | Day 0
  Number
Orexin levels in CSF in NT1 patients | Day 0
  Measured by Radio-immuno-assay (pg/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Dunyach-Remy, Principal Investigator — CHU de Nimes
Locations (2):
- France (2):
  - Nîmes University Hospital, Nîmes, Gard
  - Centre Hospitalier Universitaire de Montpellier, Montpellier